CLINICAL TRIAL: NCT04235426
Title: Platelet Rich Plasma Injection Versus Surgical and Medical Treatment of Mild-moderate Carpel Tunnel Syndrome.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dalia Salah Saif (Other)
Responsible Party: Sponsor-Investigator, Dalia Salah Saif, principle investigator, Menoufia University
Organization: Menoufia University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1472
Record Dates: First submitted 2020-01-17; First posted 2020-01-21 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Carpal Tunnel
MeSH Terms: conditions — Median Neuropathy | interventions — Anti-Inflammatory Agents, Non-Steroidal; Diclofenac; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- surgical group. (Experimental): 30 patients went to the surgical release of carpal tunnel.
  Interventions: Procedure: 30 patients went to surgical procedure
- medical group. (Experimental): 30 patients received conventional medical treatment (NSAIDs, diclofenac 150 mg/day for 2 weeks and 1500 g vitamin B 12 per day for 6 weeks) and hand support.
  Interventions: Drug: 30 patients received conventional medical treatment (NSAIDs, diclofenac 150 mg/day for 2 weeks and 1500 g vitamin B 12 per day for 6 weeks) and hand support.
- injection group. (Experimental): Thirty patients were injected in the carpal tunnel with a of single ultrasound-guided Platelet Rich Plasma (1-2 ml) injections treatments
  Interventions: Other: Injection

INTERVENTIONS:
Drug: 30 patients received conventional medical treatment (NSAIDs, diclofenac 150 mg/day for 2 weeks and 1500 g vitamin B 12 per day for 6 weeks) and hand support. — 30 patients received conventional medical treatment (NSAIDs, diclofenac 150 mg/day for 2 weeks and 1500 g vitamin B 12 per day for 6 weeks) and hand support.
  Arms: medical group.
Procedure: 30 patients went to surgical procedure — 30 patients went to surgical RELEASE OF TRANSVERSE VOLAR LIGAMENT.
  Arms: surgical group.
Other: Injection — Thirty patients were injected in the carpal tunnel with a of single ultrasound-guided Platelet Rich Plasma (1-2 ml) injections treatments
  Other Names: PRP injection.
  Arms: injection group.

SUMMARY:
to evaluate the therapeutic efficacy of single ultrasound guided Platelet Rich Plasma injection of the carpal tunnel Vs. surgical procedures and medical treatment and hand support in patients with mild-moderate carpal tunnel syndrome regarding pain relief and function improvement during a follow up period of 6 months.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) accounts for approximately 90% of peripheral entrapment neuropathy cases. Existing evidence based treatments for carpal tunnel syndrome, splinting, corticosteroid injection and surgery, are not 100% effective and alternative treatments are worth exploring .Surgery indicated in Patients with persistent numbness and pain, motor dysfunction with diminished grip or pinch grasping, or thenar eminence flattening. Empirical evidence indicates that many patients with CTS have self-limiting symptoms and respond to splinting and anti-inflammatory medications. Recently major attention has been drawn to platelet-rich plasma for its possible effects on axon regeneration and neurological recovery.

ELIGIBILITY:
Inclusion Criteria:

* patients with signs and symptoms of CTS and a confirmed diagnosis of mild and moderate CTS based on clinical and electrophysiological studies were included.

Exclusion Criteria:

1. pregnancy.
2. history of underlying metabolic diseases (such as diabetes mellitus, thyroid diseases, rheumatoid arthritis and etc.).
3. history of local corticosteroid injection in the past 3 months.
4. atrophy of thenar muscles.
5. previous carpal tunnel release surgery and evidence of concomitant neuropathy or radiculopathy.
6. Patients with autoimmune or hematologic disorders, NSAID consumption 2 days prior to injection, treatment with antiplatelet and anticoagulant agents, Hb level under 12 g/dl, and platelet count under 150,000 in ml.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
VAS (Visual Analogue Scale), | at baseline and at 3 and 6 months post injection.
  The pain severity was determined by the patients, on a scale of 0 (no pain) to 10 (agonizing pain)
Electrophysiological study of median nerve. | at baseline and at 3 and 6 months post injection.
  motor and sensory conductive of the median nerve.

CONTACTS AND LOCATIONS:
Locations (1):
- Dalia Saif, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided